CLINICAL TRIAL: NCT04229082
Title: Next Generation Probiotics (NGPs) for Metabolic Health - Metagenomic Analysis to Identify NGP Candidates Correlated With Body Weight or Metabolic Markers
Brief Title: Next Generation Probiotics (NGPs) for Metabolic Health
Status: Completed | Type: Observational
Sponsor: Danisco (Industry)
Collaborators: Oy Medfiles Ltd (Industry); 4Pharma Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MFDU002
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fecal, urine, blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lean: BMI between 18-25
  Interventions: Other: observational
- obese: BMI between 27.5-35
  Interventions: Other: observational

INTERVENTIONS:
Other: observational

SUMMARY:
To identify differences in the intestinal microbiota by metagenomics analyses between lean and obese subjects

ELIGIBILITY:
Inclusion Criteria:

1. Females.
2. Age between 20 to 50 years.
3. Obtained his/her informed consent after verbal and written information.
4. Sufficient general health and orientation for participating in the study as evaluated by the study personnel.
5. Have a high probability for compliance with and completion of the study.
6. Available for study visits and availability for food
7. Normal gastrointestinal function.
8. Willingness to provide faecal, urine and blood samples and keep food diary

Exclusion Criteria:

Lactobacillus Rhamnosus GG or reuteri, bifidobacteria enriched products) in the past 6 weeks. 12. Use of anti-obesity drugs. 13. Active or recent (last 3 months) participation in a weight loss program including weight change (increase or loss) of 3 kg during the past three months. 14. Special diets e.g. Vegetarian, Vegan, Diets with intention to use certain limited food groups only (like paleo diet, egg-grape diet etc.) 15. History of chronic active inflammatory disorders. 16. History of bariatric surgery. 17. Regular use of non-steroidal anti-inflammatory drugs, corticosteroids, or equivalent immunomodulatory drugs. 18. Ongoing or recent (last 3 months) antibiotic treatment. 19. Immunosuppression or ongoing therapy causing immunosuppression. 20. Use of vitamin supplementations beyond Recommended Daily Intake levels during the previous 2 months and during the study, except for vitamin D supplementation up to 20 μg/day.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: General adult population
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2017-06-09 (Actual)

PRIMARY OUTCOMES:
evaluate the differences in the intestinal microbiota profile between lean and obese subjects. | 1 week